CLINICAL TRIAL: NCT04280068
Title: HealthCall-S: Targeting Non-virally Suppressed Adults With Alcohol Use Disorder in HIV Primary Care
Brief Title: Targeting Non-virally Suppressed Adults With Alcohol Use Disorder in HIV Primary Care
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19 recruitment and enrollment of participants was halted
Sponsor: Research Foundation for Mental Hygiene, Inc. (Other)
Collaborators: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Deborah Hasin, Professor of Epidemiology (in Psychiatry) Columbia University, Research Foundation for Mental Hygiene, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AA023163-05
Record Dates: First submitted 2020-02-17; First posted 2020-02-21 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Alcohol Dependence; HIV/AIDS
Keywords: Human Immunodeficiency Virus; Unsafe Drinking; Antiretroviral Therapy (ART); Clinician Guide (CG)
MeSH Terms: conditions — Alcoholism; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to an evidenced-based brief behavioral intervention.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will be blinded to arms assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinician Guide (Active Comparator): Clinician Guide is an evidence-based, NIAAA-advocated approach to brief intervention for heavy drinking in primary care settings.
  Interventions: Behavioral: Clinician Guide (CG)
- Clinician Guide plus HealthCall (Active Comparator): Clinician Guide plus the use of HealthCall, a smartphone application to monitor daily alcohol use, ART adherence and other health behaviors.
  Interventions: Behavioral: Clinician Guide (CG); Behavioral: Clinician Guide plus HealthCall

INTERVENTIONS:
Behavioral: Clinician Guide (CG) — An evidence-based, intervention approach to reduce heavy drinking in primary care settings.
Behavioral: Clinician Guide plus HealthCall — HealthCall is a smartphone application designed to help participants keep track of their daily alcohol use, medication adherence and a few other health behaviors through brief daily use.
  Arms: Clinician Guide plus HealthCall

SUMMARY:
The proposed pilot study is a randomized feasibility trial of technology-enhanced brief intervention for drinking reduction and antiretroviral therapy (ART) adherence in 60 non-virally suppressed HIV participants who meet criteria for DSM-5 Alcohol Use Disorder (AUD) in a Primary Care clinic.

Study sample will be recruited from a large urban HIV primary care clinic at Montefiore Hospital where the investigators previously successfully enrolled, randomized and treated study participants

The interventions consist of brief meetings to discuss drinking and ART adherence enhanced with daily self-monitoring through the use of a smartphone application that tracks drinking and other aspects of health. These meetings will be based on the Clinician's Guide, a brief intervention for heavy drinking in primary care settings advocated by the National Institute on Alcohol Abuse and Alcoholism. Participants will be assessed at baseline, 30, 60, 90 days, and 6 months after baseline. By the end of treatment (60 days) and throughout the follow-up period, alcohol use is expected to highest among participants who receive the Clinician's Guide alone, and lowest among participants who receive the Clinician's Guide plus the smartphone application.

DETAILED DESCRIPTION:
HIV infection is a widespread health problem in the U.S. Antiretroviral (ART) therapy has increased longevity and changed the nature of risk factors for morbidity and mortality. Alcohol consumption has become an increasingly serious health issue among HIV primary care patients. Drinking is a key factor in progression to severe liver damage (especially those co-infected with hepatitis), and liver disease is now one of the most common causes of death among those with HIV. Excess drinking is also associated with medication noncompliance, reduces the effect of antiretroviral treatment, and is linked to other health problems. Therefore, helping HIV patients reduce unsafe drinking is crucial to their long-term health. This study aims to evaluate an evidence-based approach, the Clinician Guide, when combined with an innovative smartphone application designed to help users track drinking and ART adherence and other aspects of health. An effective, easily implemented alcohol-reduction intervention could be incorporated into standard care in HIV clinics to help prevent or slow the progress of some medical problems in HIV-infected individuals, improve ART medication compliance, prolong lifespan and decrease risk behavior associated with alcohol use.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Patient had 4 or more drinks on any day in prior 30 days
* Patient meets criteria for DSM5 current alcohol dependence
* HIV+
* Non-virally suppressed (HIV RNA > 200 last check)
* Able to give informed consent

Exclusion Criteria:

* Multi-drug resistant HIV and no fully suppressive treatment regimen is available
* Unwilling to take ART medications
* Patient is psychotic, suicidal, or homicidal
* Patient has gross cognitive impairment
* Patient does not speak English or Spanish
* Patient has definite plans to leave the greater New York metropolitan area within the study period
* Patient has vision/hearing impairment that would preclude participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-03-27 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Alcohol Consumption | Baseline, 30, 60 days (end-of-treatment), 3, and 6 months
  Assessing change over time in the total number of drinks in the past 30 days from baseline to each time point.

SECONDARY OUTCOMES:
Change in HIV Viral Load | Baseline and 6 months
  Assessing change in viral load count between two time points.
Change in ART medication adherence | Baseline, 30, 60 days (end-of-treatment), 3, 5 and 6 months
  Assessing change in ART medication usage between baseline and each time point.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah S Hasin, PhD, Principal Investigator — New York State Psychiatric Institute & Columbia University Medical Center
Locations (1):
- Montefiore Hospital Infectious Disease clinic, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers.